CLINICAL TRIAL: NCT05577312
Title: A Phase 1/2 Clinical Study to Evaluate the Safety and Efficacy of Single Dose Intravenous Infusion of BRL-101 in Subjects With Transfusion-Dependent β-Thalassemia
Brief Title: Safety and Efficacy Evaluation of BRL-101 in Subjects With Transfusion-Dependent β-Thalassemia
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); Xiangya Hospital of Central South University (Other); Chinese Academy of Medical Sciences (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-BRL-101
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Beta-Thalassemia
Keywords: Transfusion-Dependent β-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRL-101 (Experimental): BRL-101 (autologous CD34+ hHSPCs modified with CRISPR-Cas9 at the erythroid lineage-specific enhancer of the BCL11A gene). Subjects will receive a single infusion of BRL-101.
  Interventions: Drug: BRL-101

INTERVENTIONS:
Drug: BRL-101 — CD34 + autologous hematopoietic stem and progenitor cells edited at the BCL11A enhancer site
  Other Names: BRL-101 autologous hematopoietic stem and progenitor cells injection

SUMMARY:
This is a non-randomized, open label, multi-site, single-dose, phase 1/2 study in subjects with Transfusion-Dependent β-Thalassemia (TDT). The study will evaluate the safety and efficacy of autologous CRISPR-Cas9 modified CD34+ human hematopoietic stem and progenitor cells (hHSPCs) (BRL-101)

DETAILED DESCRIPTION:
This clinical trial is a multi-center, single-arm, single-dose, open-label study without dose escalation. The proposed dose is ≥ 3 × 106 CD34 + cells/kg administered as a single intravenous infusion. The primary objective of Phase 1 is to explore the safety of the study drug in different age groups. For subjects of each age group, myeloablative conditioning and dosing of the remaining subjects was initiated only after completion of dosing and safety observations and assessments in sentinel subjects. The Phase 2 primary objective was to determine the effectiveness of BRL-101 administered intravenously to patients with TDT.

ELIGIBILITY:
Key Inclusion Criteria:

* Fully understand and voluntarily sign informed consent. 3-35years old. At least one legal guardian and/or Subjects to sign informed consent.
* Clinically diagnosed as β-thalassemia major, phenotypes including β0β0, β+β+, β+β0, βEβ0 genotype.
* Subjects with no affection with HIV, TP, HBV, HCV, CMV and EBV.
* Subjects body condition eligible for autologous stem cell transplant.

Key Exclusion Criteria:

* Subjects acceptable for allogeneic hematopoietic stem cell transplantation and have an available fully matched related donor.
* Active bacterial, viral, or fungal infection.
* Treated with erythropoietin prior 3 months.
* Immediate family member with any known hematological tumor.
* Subjects with severe psychiatric disorders to be unable to cooperate.
* Prior hematopoietic stem cell transplant (HSCT).

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of stem cell engrafted subjects | Within 42 Days After BRL-101 Infusion
  Stem cell engraftment was defined as an absolute peripheral blood neutrophil count of ≥ 0.5 × 109/L for 3 consecutive days within 42 days following BRL-101 intravenous infusion.
Time to neutrophil engraftment | Up to 12 Months After BRL-101 Infusion
  Defined as Day 1 of absolute peripheral blood neutrophil count ≥ 0.5 × 109/L for 3 consecutive days
Frequency, severity, and relationship to BRL-101 of adverse events over 12 months following BRL-101 infusion | Up to 12 Months After BRL-101 Infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochen Wang, PhD, Study Chair — Bioray Laboratories
Locations (4):
- China (4):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No